CLINICAL TRIAL: NCT01303848
Title: Circadian Rhythm of Blood Lactate, Lipid Transferproteins and Genetic Markers (PPARs, CLOCK, Bmal1)
Brief Title: Circadian Rhythm of Blood Lactate
Status: Completed | Type: Observational
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Collaborators: State University of New York - Downstate Medical Center (Other)
Responsible Party: Principal Investigator, Axel Schlitt, PD Dr. med. habil., Martin-Luther-Universität Halle-Wittenberg
Other Study IDs: UKH2011Sport1
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
Keywords: Blood lactate; Lipid transfer proteins; Lactate; PLTP; CETP; PPARs; CLOCk; Bal1
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy probands: Healthy probands, age between 18 and 40 years
  Interventions: Other: Blood Sampling

INTERVENTIONS:
Other: Blood Sampling — Blood Sampling over 24 hours

SUMMARY:
To elucidate whether blood lactate, lipid transfer proteins and PPARs/CLOCK/Bal1 have a circadian rhythm

DETAILED DESCRIPTION:
Blood will be drawn fasting and then every hour over a period of 24 hours in 30 healthy probands.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40 years old

Exclusion Criteria:

* Inability/unwilling to give written informed consent
* Chronic disease

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 30 healthy probands
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-02; Primary Completion 2011-12 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Circadian rhythm of blood lactate | 5 months
  Blood samples

SECONDARY OUTCOMES:
Circadian rhythm of Lipid transfer proteins | 5 months
  Blood
Circadian rhythm of PPARs, CLOCK and Bal1 | 5 months
  Blood

CONTACTS AND LOCATIONS:
Overall Officials: Axel Schlitt, MD, Principal Investigator — Department of Medicine III, University Clinic Halle, Martin Luther-University Halle-Wittenberg
Locations (1):
- University Clinic Halle, Martin Luther-University Halle-Wittenberg, Halle, Germany